CLINICAL TRIAL: NCT02392910
Title: Hospitalization and Mortality in Iron Deficient, Anemic Patients With Chronic Kidney (CKD) and Heart Failure Receiving Intravenous Iron Therapy: A Five Year Follow-up From a Pilot Study
Brief Title: Hospitalization & Mortality in Patients With Iron Deficiency CKD and HF Treated With i.v. Iron.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Aleman (Other)
Responsible Party: Principal Investigator, Jorge Eduardo Toblli, Jorge Eduardo Toblli, MD; PhD; FASN. Professor of Medicine. Chief of Nephrology., Hospital Aleman
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5427-06/07
Record Dates: First submitted 2015-03-15; First posted 2015-03-19 (Estimated); Last update posted 2015-03-19 (Estimated); Status verified 2015-03

CONDITIONS: Iron Deficiency; Heart Failure; Chronic Kidney Disease
Keywords: Iron Sucrose; Mortality; Hospitalization
MeSH Terms: conditions — Iron Deficiencies; Heart Failure; Renal Insufficiency, Chronic | interventions — Ferric Oxide, Saccharated; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Other): Placebo
  Interventions: Drug: Placebo
- Group B (Other): Iron Sucrose
  Interventions: Drug: Iron Sucrose

INTERVENTIONS:
Drug: Iron Sucrose — At each visit, the patient lay on a stretcher and underwent a vein cannulation in the forearm with a commercial canula no. 16, which was connected to IV tubing that was connected to a bag contained 200 ml isotonic saline solution 0.9% plus 200 mg of Iron Sucrose. Each infusion was administered throughout 60 min. This scheme was followed for 5 consecutive weeks.
  Other Names: Venofer
  Arms: Group B
Drug: Placebo — At each visit, the patient lay on a stretcher and underwent a vein cannulation in the forearm with a commercial canula no. 16, which was connected to IV tubing that was connected to a bag of isotonic saline solution 0.9% (200 ml). Each infusion was administered throughout 60 min. This scheme was followed for 5 consecutive weeks.
  Other Names: Sodium Chloride 0.9%
  Arms: Group A

SUMMARY:
Iron deficiency, independent of anemia, appears to increase morbidity and mortality as well as impairing health-related quality of life in chronic heart failure (CHF), and these effects are compounded when patients also experience chronic kidney disease (CKD). This study was designed to determine the effects of intravenous iron treatment on morbidity and mortality following an initial 6-month period and a longer period of up to 5 years.

DETAILED DESCRIPTION:
Effect of i.v. iron sucrose on iron parameters and anemia

* During the original 6 month trial, patients in the i.v. iron group received 1000mg iron per the protocol. No patients required iron in the subsequent 6 months.
* During the subsequent follow-up, patients required a mean of between 165 and 274 mg iron per year (range: 0 to 600 mg per patient per year).
* Post the initial 1000mg iron, 19 out of 20 patients required at least a second dose of i.v. iron. Most patients required only one or two doses per year.
* The average time to requiring a second iron administration was 14.5 ± 2.7 months (range: 14 months, 23 months).
* Correction of iron deficiency (ID) resulted in statistically significant increases in transferrin saturation (TSAT) throughout the study (p < 0.01 untreated group). At all measured points, TSAT values in the treated group were at least on target (> 20% increase).
* For serum ferritin, significant differences were observed at 6 months and 1 year however this difference was not observed at 5 years post baseline where serum ferritin values were 173ng/mL and 167ng/mL for the control and IV iron groups, respectively.
* Statistically significant improvements versus the untreated group were observed for both hemoglobin (Hb) and creatinine clearance (CrCl) as well as for left ventricular ejection fraction (LVEF) and New York Heart Association (NYHA) functional class at each year.

Effect of i.v. iron sucrose on hospitalizations and mortality

* There were numerically fewer hospitalization reported at 6 months compared to those among untreated patients (0% and 25%, respectively), although the difference versus untreated patients was not statistically significant (p=ns).
* At 1 year after commencing the original study, the number of patients requiring a hospitalization (for any reason) was 50% in the control group and 10% in the IV iron group (p<0.01).
* By 5 years follow-up these rates had increased to 85% in the control arm and 20% in the IV iron treated group (p<0.01).
* In relation to all-cause mortality, there were no deaths in either group after the first 6 months. The number of deaths due to any cause after year 1 had increased in both groups (20% in the untreated group, 5% in the treated group; p=ns).
* At 5 years follow-up, 11 (55%) of patients in the control arm were deceased, compared with 4 (20%) in the IV iron treated group (p < 0.05).

ELIGIBILITY:
Inclusion:

* LV ejection fraction (EF) ≤ 35%
* New York Heart Association (NYHA) functional class II to IV
* Anemia with an iron deficit defined by Hb 12.5 g/dl for men and 11.5 g/dl for women, and some of the following: serum ferritin 100 ng/ml and/or with transferrin saturation (TSAT) 20%
* Creatinine clearance 90 ml/min.

Exclusion:

* Hemodialysis therapy
* Anemia not due to iron deficiency
* NYHA functional class I
* History of allergy to the iron supplements
* Acute bacterial infections, parasitism known in the 4 previous weeks
* Neoplasm
* Chronic digestive diseases
* Hypothyroidism
* Congenital cardiopathies
* Receiving iron supplements in the 4 previous weeks
* Receiving rhEPO in the 4 previous weeks
* History of hospitalization during the 4 weeks before enrollment into the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-03; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
mortality | 5 years

SECONDARY OUTCOMES:
Hospitalization | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Jorge E Toblli, MD; PhD, Principal Investigator — Hospital Aleman
Locations (1):
- Hospital Aleman, Buenos Aires, Buenos Aires F.D., Argentina

REFERENCES:
- [Background] Toblli JE, Lombrana A, Duarte P, Di Gennaro F. Intravenous iron reduces NT-pro-brain natriuretic peptide in anemic patients with chronic heart failure and renal insufficiency. J Am Coll Cardiol. 2007 Oct 23;50(17):1657-65. doi: 10.1016/j.jacc.2007.07.029. PMID 17950147